CLINICAL TRIAL: NCT00900757
Title: Phase II Study to Evaluate the Efficacy and Safety of Intravenous Palonosetron in Primary Glioma Patients Receiving Standard Radiotherapy and Concomitant Temozolomide
Brief Title: Intravenous Palonosetron With Radiotherapy and Concomitant Temozolomide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00015573
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2014-03

CONDITIONS: Malignant Glioma
Keywords: Primary Glioma; Palonosetron; Standard Radiotherapy; Temozolomide
MeSH Terms: conditions — Glioma | interventions — Palonosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Palonosetron (Experimental): Single Arm trial of Palonosetron for the prevention of RINV in primary malignant glioma patients receiving radiation therapy (RT) and concomitant temozolomide (TMZ)
  Interventions: Drug: Palonosetron (PALO)

INTERVENTIONS:
Drug: Palonosetron (PALO) — Eligible patients should receive a planned total dose of 54-60 GY of radiation and 75 mg/m2 of daily temozolomide for a total of six weeks of treatment. For each week of radiation patients will receive a single 0.25 mg intravenous dose of palonosetron 30 minutes before each week of radiation fraction. This schedule will be repeated for each week of radiation for a total of 6 weeks.
  Other Names: Aloxi

SUMMARY:
1. Purpose and objective:

1. To determine the safety and tolerability of palonosetron in the prevention of radiation induced nausea and vomiting (RINV) in primary glioma patients receiving radiation (RT) and concomitant temozolomide (TMZ).
2. To determine the efficacy of palonosetron in primary glioma patients receiving six weeks of RT and concomitant TMZ
3. To evaluate the effect s of palonosetron on the quality of life of primary glioma patients receiving six weeks of RT and Concomitant TMZ.

2. Study activities and Population group: We will conduct a phase II single arm trial of Palonosetron (PALO) for the prevention of RINV in primary malignant glioma patients receiving radiation therapy (RT) and concomitant temozolomide (TMZ). All eligible patients should receive a planned total dose of 54-60 GY of radiation and 75 mg/m2 of daily temozolomide for a total of six weeks of treatment. For each week of radiation patients will receive a single 0.25 mg intravenous dose of palonosetron 30 minutes before each week of radiation fraction. This schedule will be repeated for each week of radiation for a total of 6 weeks. Forty subjects with gliomas will participate.

3. Data analysis and risk/safety issues: The frequency of toxicity will be summarized by type and the most severe grade experienced. The complete response rate, defined as the proportion of patients with no emetic episode or use of rescue medication while receiving radiation and concomitant temozolomide, will be estimated with a 95% confidence interval.

DETAILED DESCRIPTION:
We will conduct a phase II single arm trial of Palonosetron (PALO) for the prevention of RINV in primary malignant glioma patients receiving radiation therapy (RT) and concomitant temozolomide (TMZ). All eligible patients should receive a planned total dose of 54-60 GY of radiation and 75 mg/m2 of daily temozolomide for a total of six weeks of treatment. For each week of radiation patients will receive a single 0.25 mg intravenous dose of palonosetron approximately 30 minutes before each week of radiation fraction. This schedule will be repeated for each week of radiation for a total of 6 weeks. After the start of radiation the type of rescue medication will be up to the investigator's discretion (however given the results of recent published phase II study by Navari et. al. we recommend using olanzapine for rescue medication). All patients will be given written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Karnofsky ≥ 60%;
* Hematocrit > 29%, absolute neutrophil count (ANC) > 1,000 cells/*1, platelets > 100,000 cells/*I;
* Serum creatinine < 1.4 mg/dl; serum glutamate oxaloacetate transaminase (SGOT) and bilirubin < 1.5 times upper limit of normal;
* For patients on corticosteroids, they must have been on a stable dose for 1 week prior to entry, and the dose should not be escalated over entry dose level, if clinically possible;
* Signed informed consent approved by the Institutional Review Board prior to patient entry;
* If sexually active, patients w8ill take contraceptive measures for the duration of the treatments.

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids;
* Inability or unwillingness to cooperate with the study procedures;
* Prophylactic medication for the prevention of nausea and vomiting 24 hours prior to the start of radiation therapy through the full course of radiation therapy is prohibited, with the exception of the study drug. Corticosteroids will be allowed for treatment of cerebral swelling. Rescue medication for treatment of nausea and vomiting is permitted after radiation therapy at the discretion of the investigator. The agent, dose, and time of administration will be recorded in the patient diary;
* Previous participation in any clinical trial involving palonosetron;
* Any vomiting, retching, or NCI Common Toxicity Criteria version 3.0 grade 2-4 nausea in the 24 hours preceding radiation and chemotherapy;
* Ongoing vomiting from any organic etiology;
* Will receive radiotherapy of upper abdomen within one week prior to or during the study;
* Received palonosetron within 14 days prior to study enrollment;
* Prior and Concomitant Medications for Prevention/Treatment of Nausea and Vomiting;
* Prior and Concomitant Cancer Chemotherapy and Radiotherapy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Lou Affronti, RN, MSN, ANP, Principal Investigator — Duke Health
Locations (1):
- The Preston Robert Tisch Brain Tumor Center at Duke, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Palonosetron
Started | 57
Completed | 38
Not Completed | 19
Not completed — screen failure | 19

BASELINE CHARACTERISTICS:
Arm/Group | Palonosetron
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Palonosetron as Determined by the Number of Participants Who Experience Unacceptable Toxicity
Description: The number of participants with unacceptable toxicity defined as ≥grade 3, non-hematologic toxicities that are possibly, probably or definitely related to the study regimen.
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Palonosetron
Number analyzed (Participants) | 38
participants | 5

2. Secondary Outcome: Complete Response
Description: The percentage of participants with a complete response defined as no emetic episode or use of rescue medication while receiving radiation (XRT) and concomitant temozolomide (TMZ).
Time Frame: 6 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Palonosetron
Number analyzed (Participants) | 38
percentage of participants
  Week 1 of XRT and TMZ (n=38) | 74 [57 to 87]
  Week 2 of XRT and TMZ (n=38) | 79 [63 to 90]
  Week 3 of XRT and TMZ (n=38) | 76 [60 to 89]
  Week 4 of XRT and TMZ (n=38) | 74 [57 to 87]
  Week 5 of XRT and TMZ (n=36) | 67 [49 to 81]
  Week 6 of XRT and TMZ (n=34) | 71 [53 to 85]
  Overall (across weeks 1-6 of XRT and TMZ) (N=34) | 44 [27 to 62]

3. Secondary Outcome: Change in the Functional Living Index - Emesis (FLIE) Score From Baseline to Each Week of Radiation (XRT) and Temozolomide (TMZ) Treatment
Description: The FLIE is a 18-item validated questionnaire for assessing the effects of chemotherapy-induced nausea and emesis on quality of life and daily functioning. The raw score range is 18-126 with higher scores indicating better quality of life. For each week of XRT and TMZ, the change from baseline was calculated by subtracting the baseline score from the mean of the day 1, 3 and 6 scores. A negative change represents worsening in quality of life due to nausea and emesis.
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Palonosetron
Number analyzed (Participants) | 38
units on a scale
  Week 1 of XRT and TMZ (n=38) | -3.3 [-6.8 to 0.2]
  Week 2 of XRT and TMZ (n=38) | -2.7 [-5.9 to 0.4]
  Week 3 of XRT and TMZ (n=38) | -1.9 [-4.1 to 0.3]
  Week 4 of XRT and TMZ (n=38) | -3.9 [-8.1 to 0.3]
  Week 5 of XRT and TMZ (n=36) | -5.5 [-11.0 to -0.1]
  Week 6 of XRT and TMZ (n=34) | -4.1 [-7.5 to -0.7]

4. Secondary Outcome: Percentage of Participants With a Osoba Nausea Module Maximum Standardized Score of Zero for Each Week of Radiation (XRT) and Temozolomide (TMZ)
Description: Percentage of participants with a Osoba nausea module maximum standardized score of zero for each week of radiation (XRT) and Temozolomide (TMZ). The Osoba nausea module is a 5-item questionnaire assessing the effect of nausea on quality of life and daily functioning. Raw scores range from 5-20 and have been converted to standardized scores (0-100) using the formula: std_score = round((raw_score - 5) * 6.66). Lower scores indicate better quality fo life. The maximum standardized score of all nausea scores collected during the week (days 1, 3 and 6) was used for this outcome.
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Palonosetron
Number analyzed (Participants) | 38
percentage of participants
  Week 1 of XRT and TMZ (n=38) | 76
  Week 2 of XRT and TMZ (n=38) | 79
  Week 3 of XRT and TMZ (n=38) | 79
  Week 4 of XRT and TMZ (n=38) | 79
  Week 5 of XRT and TMZ (n=35) | 71
  Week 6 of XRT and TMZ (n=34) | 79

5. Secondary Outcome: Percentage of Participants With a Osoba Vomiting/Retching Module Maximum Standardized Score of Zero for Each Week of Radiation (XRT) and Temozolomide (TMZ)
Description: Percentage of participants with a Osoba vomiting/retching module maximum standardized score of zero for each week of radiation (XRT) and Temozolomide (TMZ). The Osoba vomiting/retching module is a 5-item questionnaire assessing the effect of vomiting/retching on quality of life and daily functioning. Raw scores range from 5-20 and have been converted to standardized scores (0-100) using the formula: std_score = round((raw_score - 5) * 6.66). Lower scores indicate better quality fo life. The maximum standardized score of all vomiting/retching scores collected during the week (days 1, 3 and 6) was used for this outcome.
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Palonosetron
Number analyzed (Participants) | 38
percentage of participants
  Week 1 of XRT and TMZ (n=38) | 87
  Week 2 of XRT and TMZ (n=38) | 89
  Week 3 of XRT and TMZ (n=38) | 100
  Week 4 of XRT and TMZ (n=38) | 92
  Week 5 of XRT and TMZ (n=35) | 89
  Week 6 of XRT and TMZ (n=34) | 97

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: The adverse events for this study were collected using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, and have been converted to CTCAE version 4.0 for entry into ClinicalTrials.gov.
Arm/Group | Palonosetron
Serious Adverse Events (participants affected / at risk) | 5/38
Other Adverse Events (participants affected / at risk) | 36/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palonosetron (N=38)
Atrial fibrillation (Cardiac disorders) | 1
Edema face (General disorders) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palonosetron (N=38)
Anemia (Blood and lymphatic system disorders) | 2
Blurred vision (Eye disorders) | 15
Constipation (Gastrointestinal disorders) | 21
Diarrhea (Gastrointestinal disorders) | 8
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 9
Edema limbs (General disorders) | 3
Fatigue (General disorders) | 21
Fever (General disorders) | 2
Infections and infestations - Other, specify (Infections and infestations) | 11
Wound infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 2
Investigations - Other, specify (Investigations) | 1
Platelet count decreased (Investigations) | 6
Weight loss (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 12
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 4
Ataxia (Nervous system disorders) | 11
Cognitive disturbance (Nervous system disorders) | 16
Depressed level of consciousness (Nervous system disorders) | 15
Dizziness (Nervous system disorders) | 13
Dysphasia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 19
Memory impairment (Nervous system disorders) | 15
Peripheral motor neuropathy (Nervous system disorders) | 15
Peripheral sensory neuropathy (Nervous system disorders) | 8
Seizure (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 5
Confusion (Psychiatric disorders) | 14
Depression (Psychiatric disorders) | 18
Insomnia (Psychiatric disorders) | 17
Urinary incontinence (Renal and urinary disorders) | 6
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Rash acneiform (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution will provide Eisai with a copy of any manuscript, paper, or poster connected with the study at least 30 days prior to submission to journal/presentation in order for Eisai to review for Eisai's Confidential Information (CI). Should Eisai notify Institution with such 30 day period that materials contain CI, Institution agrees to delay submission/publication/presentation for an additional 60 days to allow Eisai to seek patent or other protection.